CLINICAL TRIAL: NCT02345070
Title: Efficacy and Safety of SAR156597 in the Treatment of Idiopathic Pulmonary Fibrosis (IPF): A Randomized, Double-blind, Placebo-controlled, 52-week Dose-ranging Study
Brief Title: Efficacy and Safety of SAR156597 in the Treatment of Idiopathic Pulmonary Fibrosis
Acronym: ESTAIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI11772; 2014-003933-24 (EudraCT Number); U1111-1154-6083 (Other: UTN)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo qw (Placebo Comparator): Participants received one injection of placebo (matched to SAR156597) subcutaneously once every week (qw) for 52 weeks.
  Interventions: Drug: placebo
- SAR156597 200 mg q2w (Experimental): Participants received one injection of SAR156597 200 mg subcutaneously once every 2 weeks (q2w) alternating with placebo (matched to SAR156597) for 52 weeks.
  Interventions: Drug: SAR156597; Drug: placebo
- SAR156597 200 mg qw (Experimental): Participants received one injection of SAR156597 200 mg subcutaneously qw for 52 weeks.
  Interventions: Drug: SAR156597

INTERVENTIONS:
Drug: SAR156597 — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: SAR156597 200 mg q2w; SAR156597 200 mg qw
Drug: placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo qw; SAR156597 200 mg q2w

SUMMARY:
Primary Objective:

To evaluate, in comparison with placebo, the efficacy of 2 dose levels/regimens of SAR156597 administered subcutaneously during 52 weeks on lung function of participants with Idiopathic Pulmonary Fibrosis (IPF).

Secondary Objectives:

To evaluate the efficacy of 2 dose levels/regimens of SAR156597 compared to placebo on IPF disease progression.

To evaluate the safety of 2 dose levels/regimens of SAR156597 compared to placebo in participants with IPF.

DETAILED DESCRIPTION:
The total study duration of study was expected up to 68 weeks (screening period of 4 weeks, treatment period of 52 weeks, and 12 weeks of follow up).

ELIGIBILITY:
Inclusion criteria :

* Adult male or female participants.
* Documented diagnosis of IPF according to the current 2011 American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/ American Latin Thoracic Association (ATS/ERS/JRS/ALAT) guidelines.
* Signed written informed consent.

Exclusion criteria:

* Age less than or equal to 40 years.
* IPF disease diagnosis greater than 5 years.
* Forced vital capacity (FVC) less than (<) 40 percent (%) of predicted value.
* Carbon monoxide diffusing lung capacity (DLCO) corrected for hemoglobin <30% of predicted value.
* Severe chronic obstructive bronchitis as characterized by forced expiratory volume in 1 second /forced vital capacity (FEV1/FVC) <0.70.
* Need for 24 hours of oxygen therapy or oxygen saturation <88% after 10 minutes breathing ambient air at rest.
* Known diagnosis of significant respiratory disorders other than IPF.
* Pulmonary artery hypertension requiring a specific treatment.
* Currently listed and/or anticipated for lung transplantation within the next 6 months (on an active list).
* History of vasculitis or connective tissue disorders.
* Known human immunodeficiency virus or chronic viral hepatitis.
* Participants with active tuberculosis or incompletely treated latent tuberculosis infection.
* Use of any cytotoxic/immunosuppressive agent including but not limited to azathioprine, cyclophosphamide, methotrexate, and cyclosporine within 4 weeks prior to screening.
* Use of any cytokine modulators (etanercept, adalimumab, efalizumab, infliximab, golimumab, certolizumab, rituximab) within 12 weeks or 5 half-lives of screening (24 weeks for rituximab and 24 months for alefacept).
* Use of any investigational drug within 1 month of screening, or 5 half-lives, if known ( whichever was longer), or within 12 weeks for stem cell therapy.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (101):
- United States (18):
  - Investigational Site Number 840003, Phoenix, Arizona
  - Investigational Site Number 840020, Jacksonville, Florida
  - Investigational Site Number 840022, Loxahatchee Groves, Florida
  - Investigational Site Number 840017, Atlanta, Georgia
  - Investigational Site Number 840008, Decatur, Georgia
  - Investigational Site Number 840010, Louisville, Kentucky
  - Investigational Site Number 840009, Minneapolis, Minnesota
  - Investigational Site Number 840006, Rochester, Minnesota
  - Investigational Site Number 840026, Chesterfield, Missouri
  - Investigational Site Number 840001, Lebanon, New Hampshire
  - Investigational Site Number 840002, Summit, New Jersey
  - Investigational Site Number 840015, Jamaica, New York
  - Investigational Site Number 840023, Mineola, New York
  - Investigational Site Number 840012, New York, New York
  - Investigational Site Number 840013, Stony Brook, New York
  - Investigational Site Number 840014, Philadelphia, Pennsylvania
  - Investigational Site Number 840011, Dallas, Texas
  - Investigational Site Number 840024, Everett, Washington
- Argentina (6):
  - Investigational Site Number 032009, Caba
  - Investigational Site Number 032005, Caba
  - Investigational Site Number 032001, La Plata
  - Investigational Site Number 032004, Mendoza
  - Investigational Site Number 032002, San Miguel de Tucumán
  - Investigational Site Number 032007, Vicente López
- Australia (5):
  - Investigational Site Number 036005, Camperdown
  - Investigational Site Number 036004, Darlinghurst
  - Investigational Site Number 036002, Frankston
  - Investigational Site Number 036003, Murdoch
  - Investigational Site Number 036001, Nundah
- Canada (2):
  - Investigational Site Number 124003, Toronto
  - Investigational Site Number 124002, Vancouver
- Chile (6):
  - Investigational Site Number 152003, Quillota
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152006, Santiago
  - Investigational Site Number 152002, Talca
  - Investigational Site Number 152007, Viña del Mar
- Colombia (3):
  - Investigational Site Number 170004, Armenia
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170005, Cali
- Czechia (4):
  - Investigational Site Number 203002, Hradec Králové
  - Investigational Site Number 203004, Olomouc
  - Investigational Site Number 203003, Prague
  - Investigational Site Number 203001, Prague
- Denmark (2):
  - Investigational Site Number 208002, Aarhus C
  - Investigational Site Number 208001, Hellerup
- France (9):
  - Investigational Site Number 250007, Bobigny
  - Investigational Site Number 250002, Lille
  - Investigational Site Number 250001, Lyon
  - Investigational Site Number 250009, Marseille
  - Investigational Site Number 250005, Montpellier
  - Investigational Site Number 250004, Nice
  - Investigational Site Number 250006, Paris
  - Investigational Site Number 250008, Toulouse
  - Investigational Site Number 250003, Tours
- Germany (5):
  - Investigational Site Number 276003, Coswig
  - Investigational Site Number 276002, Donaustauf
  - Investigational Site Number 276004, Giessen
  - Investigational Site Number 276005, Hanover
  - Investigational Site Number 276001, Heidelberg
- Investigational Site Number 300001, Heraklion, Greece
- Israel (5):
  - Investigational Site Number 376001, Haifa
  - Investigational Site Number 376004, Kfar Saba
  - Investigational Site Number 376002, Petah Tikva
  - Investigational Site Number 376005, Rehovot
  - Investigational Site Number 376003, Tel Litwinsky
- Italy (6):
  - Investigational Site Number 380003, Catania
  - Investigational Site Number 380001, Forlì
  - Investigational Site Number 380005, Milan
  - Investigational Site Number 380002, Orbassano
  - Investigational Site Number 380006, Pisa
  - Investigational Site Number 380004, Siena
- Mexico (4):
  - Investigational Site Number 484002, Mexico City
  - Investigational Site Number 484001, Monterrey
  - Investigational Site Number 484005, Monterrey
  - Investigational Site Number 484003, San Juan del Río
- Portugal (2):
  - Investigational Site Number 620003, Porto
  - Investigational Site Number 620004, Vila Nova de Gaia
- South Korea (6):
  - Investigational Site Number 410005, Bucheon-si
  - Investigational Site Number 410001, Incheon
  - Investigational Site Number 410006, Seongnam
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410004, Seoul
- Spain (7):
  - Investigational Site Number 724003, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724001, L'Hospitalet de Llobregat
  - Investigational Site Number 724004, Lugo
  - Investigational Site Number 724006, Majadahonda
  - Investigational Site Number 724005, Palma de Mallorca
  - Investigational Site Number 724007, Sabadell
- Turkey (Türkiye) (6):
  - Investigational Site Number 792005, Ankara
  - Investigational Site Number 792006, Istanbul
  - Investigational Site Number 792001, Istanbul
  - Investigational Site Number 792004, Istanbul
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792002, Izmir
- United Kingdom (4):
  - Investigational Site Number 826002, Cambridge
  - Investigational Site Number 826003, Exeter
  - Investigational Site Number 826004, Leicester
  - Investigational Site Number 826001, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 101 active centers in 19 countries. A total of 652 participants were screened between May 2015 and May 2016, of whom, 327 participants were randomized in 1:1:1 ratio to placebo: SAR156597 200 milligram (mg) once every 2 weeks (q2w): SAR156597 200 mg once every week (qw).
Pre-assignment Details: Participants were stratified at the moment of randomization according to background therapy (participants with background anti-fibrotic therapy with either pirfenidone or nintedanib versus participants without background anti-fibrotic therapy).
Groups:
- Placebo qw: Participants received one injection of placebo (matched to SAR156597) subcutaneously qw for 52 weeks.
- SAR156597 200mg q2w: Participants received one injection of SAR156597 200 mg subcutaneously q2w alternating with placebo (matched to SAR156597) for 52 weeks.
- SAR156597 200mg qw: Participants received one injection of SAR156597 200 mg subcutaneously qw for 52 weeks.
Period: Overall Study
Arm/Group | Placebo qw | SAR156597 200mg q2w | SAR156597 200mg qw
Started (Randomized) | 110 | 109 | 108
Treated | 109 | 108 | 108
Completed | 90 | 98 | 85
Not Completed | 20 | 11 | 23
Not completed — Adverse Event | 12 | 8 | 16
Not completed — Poor compliance to protocol | 2 | 0 | 0
Not completed — Other than specified above | 6 | 3 | 7

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo qw | SAR156597 200mg q2w | SAR156597 200mg qw | Total
Number analyzed (Participants) | 110 | 109 | 108 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.6) | 67.4 (7.2) | 68.0 (7.6) | 68.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 32 | 27 | 81
  Male | 88 | 77 | 81 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 105 | 104 | 99 | 308
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 52
Description: FVC is a standard pulmonary function parameter measured by spirometry and used to quantify respiratory capacity (inspiration and expiration). It is a widely used objective measure of disease status in participants with Idiopathic Pulmonary Fibrosis (IPF). The primary variable was recorded as percent (%) of predicted value, which takes into account the height, gender, and age of the participant. The outcome measure measured the change in lung function from baseline at week 52.
Time Frame: Baseline, Week 52
Population: Modified intent-to-treat (mITT) population: All participants who received at least 1 study injection, had valid baseline percent predicted FVC measurement, and had at least 1 post-baseline percent predicted FVC measurement. Here, 'Overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent predicted FVC
Arm/Group | Placebo qw | SAR156597 200mg q2w | SAR156597 200mg qw
Number analyzed (Participants) | 81 | 89 | 75
percent predicted FVC | -5.81 (0.74) | -5.24 (0.73) | -6.31 (0.75)
Statistical Analysis 1: Comparison: Placebo qw vs SAR156597 200mg qw; A hierarchical testing procedure was used to control type I error. Testing was done sequentially in order the outcome measures were reported. Analyzed using Mixed Model for Repeated Measurements (MMRM) with fixed categorical effects of treatment arm, stratification factor (with/without background therapy), time point, treatment-by-time point interaction, stratification factor-by-treatment-by-time point interaction, and continuous fixed covariate of percent predicted FVC baseline; Test type: Superiority — The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; p = 0.6339, Mixed Models Analysis — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -0.5, 95% CI 2-sided [-2.56 to 1.56], Standard Error of Mean 1.05 — SAR156597 200mg qw versus Placebo qw
Statistical Analysis 2: Comparison: Placebo qw vs SAR156597 200mg q2w; A hierarchical testing procedure was used to control type I error. Testing was performed sequentially in the order outcome measures were reported (q2w dose group compared to placebo). Analysis was performed using MMRM with fixed categorical effects of treatment arm, stratification factor (with/without background therapy), time point, treatment-by-time point interaction, stratification factor-by-treatment-by-time point interaction, and continuous fixed covariate of percent predicted FVC baseline; Test type: Superiority — The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; p = 0.5874, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 0.56, 95% CI 2-sided [-1.47 to 2.6], Standard Error of Mean 1.04 — SAR156597 200mg q2w versus Placebo qw

2. Secondary Outcome: Time to Disease Progression: Kaplan-Meier Estimates of Probability of Disease Progression at Week 52
Description: Disease progression was defined as the time from randomization to the first occurrence of any of the following events: decrease in absolute percent predicted FVC greater than or equal to (>=) 10%, decrease in absolute percent predicted Carbon monoxide diffusing lung capacity >=15%, lung transplant, or death. The median time to disease progression was not estimated because the number of occurrence of events was too low in the SAR156597 200 mg arms.
Time Frame: From randomization to disease progression (up to Week 52)
Population: Analysis was performed on mITT population.
Measure: Number; unit: probability of disease progression
Arm/Group | Placebo qw | SAR156597 200mg q2w | SAR156597 200mg qw
Number analyzed (Participants) | 109 | 108 | 108
probability of disease progression | 0.512 | 0.460 | 0.537

3. Secondary Outcome: Time to Event: Kaplan-Meier Estimates of Probability of All Cause Mortality (Deaths) at Week 52
Description: All-cause mortality was considered for this outcome measure which was defined as the time from randomization to the date of death. The median time to event was not estimated because the number of all cause mortality was too low in the SAR156597 200 mg arms.
Time Frame: From randomization up to Week 52
Population: Analysis was performed on mITT population.
Measure: Number; unit: probability of deaths
Arm/Group | Placebo qw | SAR156597 200mg q2w | SAR156597 200mg qw
Number analyzed (Participants) | 109 | 108 | 108
probability of deaths | 0.09 | 0.08 | 0.13

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the end of follow up visit (Week 64) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported AEs and death were treatment-emergent AEs that developed/worsened and deaths that occurred during 'treatment emergent period'. Treatment period was defined as the time from the first administration of IMP to the last administration of IMP + 84 days (i.e., Week 64). Analysis was performed on safety population which included participants who received at least 1 dose or part of a dose of IMP and were analyzed according to the treatment actually received.
Arm/Group | Placebo qw | SAR156597 200mg q2w | SAR156597 200mg qw
All-Cause Mortality (participants affected / at risk) | 9/109 | 6/108 | 13/108
Serious Adverse Events (participants affected / at risk) | 26/109 | 27/108 | 46/108
Other Adverse Events (participants affected / at risk) | 81/109 | 86/108 | 79/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo qw (N=109) | SAR156597 200mg q2w (N=108) | SAR156597 200mg qw (N=108)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 2
Acute right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 2
Hepatic mass (Hepatobiliary disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 8
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
T-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Postresuscitation encephalopathy (Nervous system disorders) | 0 | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Assisted suicide (Psychiatric disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 22
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo qw (N=109) | SAR156597 200mg q2w (N=108) | SAR156597 200mg qw (N=108)
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 16 | 23 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 6 | 0
Nausea (Gastrointestinal disorders) | 9 | 9 | 9
Vomiting (Gastrointestinal disorders) | 6 | 8 | 6
Asthenia (General disorders) | 6 | 4 | 3
Injection site erythema (General disorders) | 3 | 7 | 10
Injection site haematoma (General disorders) | 2 | 5 | 6
Injection site reaction (General disorders) | 6 | 11 | 10
Pyrexia (General disorders) | 8 | 1 | 0
Bronchitis (Infections and infestations) | 12 | 18 | 10
Lower respiratory tract infection (Infections and infestations) | 2 | 11 | 6
Respiratory tract infection (Infections and infestations) | 7 | 5 | 3
Rhinitis (Infections and infestations) | 1 | 8 | 2
Upper respiratory tract infection (Infections and infestations) | 13 | 10 | 8
Urinary tract infection (Infections and infestations) | 6 | 4 | 7
Viral upper respiratory tract infection (Infections and infestations) | 15 | 18 | 12
Weight decreased (Investigations) | 9 | 9 | 8
Decreased appetite (Metabolism and nutrition disorders) | 1 | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 13 | 9
Headache (Nervous system disorders) | 7 | 5 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 22 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 13
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2015-07-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT02345070/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT02345070/SAP_001.pdf